CLINICAL TRIAL: NCT06640374
Title: Role of Clinical Pulmonary Infection Score and Sonopulmonary Infection Score in Diagnosis and Predicting Outcome of VAP in RUCU
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa khaled, Role of Clinical Pulmonary Infection Score and sonopulmonary infection score in diagnosis and Predicting Outcome of VAP in RICU Patients, Assiut University
Other Study IDs: Assiit University
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Patients with VAP in RICU Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
-Pneumonia is a bacterial, viral or fungal infection of the lungs, which causes the alveoli of the lungs to fill up with microorganisms, fluid and inflammatory cells, preventing the lungs from functioning effectively

The classification scheme for pneumonia in UK NHS hospitals is based on the setting in which the infection was mostly likely acquired:

community-acquired pneumonia (CAP), when a patient is in the hospital <48h before the pneumonia is suspected; hospital-acquired pneumonia (HAP), when a patient is in the hospital >48h before the pneumonia develops, but is not associated with mechanical ventilation; and ventilator-associated pneumonia (VAP), when a patient is mechanically ventilated and intubated for >48h before the pneumonia develops The causative pathogens in each scenario are different, and treatment strategies vary as a consequence.

DETAILED DESCRIPTION:
-Pneumonia is a bacterial, viral or fungal infection of the lungs, which causes the alveoli of the lungs to fill up with microorganisms, fluid and inflammatory cells, preventing the lungs from functioning effectively

The classification scheme for pneumonia in UK NHS hospitals is based on the setting in which the infection was mostly likely acquired:

community-acquired pneumonia (CAP), when a patient is in the hospital <48h before the pneumonia is suspected; hospital-acquired pneumonia (HAP), when a patient is in the hospital >48h before the pneumonia develops, but is not associated with mechanical ventilation; and ventilator-associated pneumonia (VAP), when a patient is mechanically ventilated and intubated for >48h before the pneumonia develops The causative pathogens in each scenario are different, and treatment strategies vary as a consequence.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 yrs or more Mechanically ventilated patients after 48 hrs after admission of ICU

Exclusion Criteria:

* Patient less than 18 yrs Patients diagnosed as pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with VAP Patients who don't develop VAP
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-09-19 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Role of Clinical Pulmonary Infection Score and sonopulmonary infection score in diagnosis of VAP and Predicting Outcome in RICU Patients | 4 years
  Diagnosis of VAP in RICU Patients

SECONDARY OUTCOMES:
Role of Clinical Pulmonary Infection Score and sonopulmonary infection score in diagnosis of VAP and Predicting Outcome in RICU Patients | 4 years
  Diagnosis of VAP in RICU PATIENTS

REFERENCES:
- [Background] Reissig A, Copetti R, Kroegel C. Current role of emergency ultrasound of the chest. Crit Care Med. 2011 Apr;39(4):839-45. doi: 10.1097/CCM.0b013e318206d6b8. PMID 21263325
- [Background] Naranje P, Bhalla AS, Sherwani P. Chest Tuberculosis in Children. Indian J Pediatr. 2019 May;86(5):448-458. doi: 10.1007/s12098-018-02847-7. Epub 2019 Feb 14. PMID 30762202